CLINICAL TRIAL: NCT03400995
Title: An Open Label, Single-dose, Single-period Study Designed to Assess the Mass Balance Recovery, Metabolite Profile and Metabolite Identification of [14C]-AK0529 in Healthy Male Subjects
Brief Title: A Study to Evaluate the Pharmacokinetics, Metabolism, and Excretion of AK0529
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Ark Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AK0529-4001
Record Dates: First submitted 2018-01-10; First posted 2018-01-17 (Actual); Last update posted 2018-09-11 (Actual); Status verified 2018-09

CONDITIONS: Healthy
MeSH Terms: interventions — ziresovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Arm (Experimental): Each subject will receive a single oral administration of a solution containing 300 mg radiolabeled AK0529 in the fasted state.
  Interventions: Drug: AK0529

INTERVENTIONS:
Drug: AK0529 — A solution containing 300 mg radiolabelled AK0529.

SUMMARY:
This phase I study is to assess the mass balance recovery after a single oral dose of [14C]-AK0529 in healthy male subjects.

DETAILED DESCRIPTION:
This is a single centre, single-dose, non-randomised, open label study. The primary objectives of this study are to assess the mass balance recovery and provide biosamples for metabolite profiling and structural identification after a single oral dose of [14C]-AK0529 in healthy male subjects. 7 subjects will be recruited to receive a single oral administration of a solution containing 300 mg AK0529. The total duration of the study will be approximately 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males
* Aged between 30 and 55 years of age, inclusive
* Body mass index of 18.0 to 35.0 kg/m2, inclusive, or, if outside the range, considered not clinically significant by the investigator and the medical monitor
* Must be willing and able to communicate and participate in the whole study
* Must have regular daily bowel movements
* Must provide written informed consent
* Must agree to use an adequate method of contraception

Exclusion Criteria:

* Subjects who have received any IMP in a clinical research study within the previous 3 months
* Subjects who are study site or sponsor employees, or immediate family members of a study site or sponsor employee
* Subjects who have previously been enrolled in this study
* History of any drug or alcohol abuse in the past 2 years
* Regular alcohol consumption >21 units per week
* Current smokers and those who have smoked within the last 12 months
* Current users of e-cigarettes and nicotine replacement products and those who have used these products within the last 12 months
* Radiation exposure. No occupationally exposed worker, as defined in the Ionising Radiation Regulations 1999, shall participate in the study
* Subjects who do not have suitable veins for multiple venepunctures/cannulation as assessed by the investigator at screening
* Abnormal liver function as assessed by clinical chemistry
* Positive drugs of abuse test result
* Positive HBsAg, HCV Ab or HIV results
* Evidence of renal impairment at screening
* History of clinically significant cardiovascular, renal, hepatic, chronic respiratory, neurological, dermatological or GI disease, or psychiatric disorder, as judged by the investigator
* Any abnormality of ECG parameters
* Any abnormality of cardiac rhythm or history thereof
* Serious adverse reaction or serious hypersensitivity to any drug or the formulation excipients
* Presence or history of clinically significant allergy requiring treatment, as judged by the investigator. Hayfever is allowed, unless it is active at screening or admission
* Donation or loss of greater than 400 mL of blood within the previous 3 months
* Subjects who are taking, or have taken, any prescribed or over-the-counter drug or herbal or any other 'alternative' remedies in the 14 days before IMP administration
* Failure to satisfy the investigator of fitness to participate for any other reason

Ages: 30 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2018-01-05 (Actual); Primary Completion 2018-02-27 (Actual); Study Completion 2018-08-30 (Actual)

PRIMARY OUTCOMES:
Amount excreted (Ae) | At approximately 6 weeks
  The amount of total radioactivity eliminated.
Percentage of the administered dose (%Ae) | At approximately 6 weeks
  The amount of total radioactivity eliminated expressed as a percentage of the dose administered.
Cumulative recovery (CumAe) | At approximately 6 weeks
  The cumulative amount of total radioactivity eliminated.
Percentage of cumulative recovery of the administered dose (Cum%Ae) | At approximately 6 weeks
  The cumulative amount of total radioactivity eliminated expressed as a percentage of the dose administered.

SECONDARY OUTCOMES:
Percentage of Subjects with Adverse Events (AEs) | From baseline up to approximately 6 weeks
  An adverse event can be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product.

CONTACTS AND LOCATIONS:
Overall Officials: ArkBio Clinical Trial, Study Director — info@arkbiosciences.com
Locations (1):
- Quotient Clinical, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No